CLINICAL TRIAL: NCT00666419
Title: Prevalence of Back Pain and Associated Risk Factors in 10-12 Year Old Schoolchildren
Status: Withdrawn | Type: Observational
Why Stopped: Recruiting at schools was slower than planned. Missing data higher than acceptable.
Sponsor: Kovacs Foundation (Other)
Collaborators: Universitat de les Illes Balears (Other)
Responsible Party: Principal Investigator, Francisco M. Kovacs, Director Spanish Back Pain Research Network (REIDE), Kovacs Foundation
Other Study IDs: FK-UIB-23
Record Dates: First submitted 2008-04-23; First posted 2008-04-24 (Estimated); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Low Back Pain
Keywords: nonspecific low back pain; schoolchildren; prevalence
MeSH Terms: conditions — Low Back Pain | interventions — Weights and Measures

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Measurement, weight, and muscle strength test — 10-12 year old schoolchildren will be weighed, measured for height, and tested for strength of their abdominal and paravertebral muscles

SUMMARY:
A large study in Mallorca, Spain showed that nonspecific low back pain is quite prevalent in adolescents 13-15 years of age (Kovacs, 2003). Since below the age of seven years hardly any child has suffered low back pain, the purpose of this study is to determine the prevalence of low back pain in children 10-12 years of age, and to investigate the risk factors associated with its occurrence.

ELIGIBILITY:
Inclusion Criteria:

* Schoolchildren born in the years 1993, 1994 or 1995
* Attending schools (public, concerted or private) in Mallorca
* Can read and write Spanish

Exclusion Criteria:

* Nor attending class on the days when the study is being done

Ages: 10 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: All 10-12 year old schoolchildren on the island of Mallorca, Spain
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2006-09; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francisco M Kovacs, MD, PhD, Study Director — Kovacs Foundation, Palma de Mallorca, 07012, Spain; Pere Palou, PhD, Principal Investigator — Universitat de les Illes Balears, Palma de Mallorca, Spain
Locations (1):
- Kovacs Foundation, Palma de Mallorca, Balearic Islands, Spain

REFERENCES:
- [Background] Balague F, Troussier B, Salminen JJ. Non-specific low back pain in children and adolescents: risk factors. Eur Spine J. 1999;8(6):429-38. doi: 10.1007/s005860050201. PMID 10664299
- [Background] Kovacs FM, Gestoso M, Gil Del Real MT, Lopez J, Mufraggi N, Ignacio Mendez J. Risk factors for non-specific low back pain in schoolchildren and their parents: a population based study. Pain. 2003 Jun;103(3):259-268. doi: 10.1016/S0304-3959(02)00454-2. PMID 12791432
- [Background] Gil del RealMT, Kovacs FM, Gestoso M, Mufraggi N, Diéguez JM. Evaluation of two questionnaires to determine exposure to risk factors for non-specific low back pain in Mallorcan schoolchildren and their parents. European Journal of Public Health 9(3): 194-199, 1999.